CLINICAL TRIAL: NCT01971385
Title: A Clinical Trial to Test the Safety and Efficacy of Squaric Acid Dibutyl Ester for the Treatment of Herpes Labialis
Brief Title: Safety and Efficacy of Squaric Acid Dibutyl Ester for the Treatment of Herpes Labialis
Acronym: Squarex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alexandra Kimball, Director, Clinical Unit for Research Trials in Skin, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013P001028
Record Dates: First submitted 2013-10-17; First posted 2013-10-29 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-05

CONDITIONS: Herpes Labialis
MeSH Terms: conditions — Herpes Labialis | interventions — squaric acid dibutyl ester

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2% Squaric Acid Sensitization (Active Comparator): 2% Squaric Acid solution will be applied for sensitization to the inner arm.
  Interventions: Drug: Squaric Acid solution
- Placebo Solution (Placebo Comparator): Patients in placebo group will be given dimethyl sulfoxide.
  Interventions: Drug: Placebo solution

INTERVENTIONS:
Drug: Squaric Acid solution
  Other Names: Squaric Acid Dibutyl Ester solution; SADBE
  Arms: 2% Squaric Acid Sensitization
Drug: Placebo solution
  Arms: Placebo Solution

SUMMARY:
Subjects with a history of recurrent herpes labialis will be sensitized with either 2% SADBE or placebo. Following this, subjects sensitized with 2% SADBE will received.2% sqauric acid or.5% squaric acid on their cold sore within 72 hours of a recurrence. Subjects sensitized with placebo solution will receive placebo solution on their cold sore within 72 hours of a recurrence. Subjects will be followed for up to 6 mos after application of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* With clinical diagnosis of herpes labialis.
* who self report having six or more episodes of herpes labialis in the previous 12 months.

Exclusion Criteria:

* Pregnant or lactating females.
* Current or recurrent infection or any underlying condition that may predispose to infection or anyone who has been admitted to the hospital due to bacteremia, pneumonia or any other serious infection.
* Therapy with glucocorticoid or immunosuppressant at time of recruitment or within past 4 weeks, except for inhaled corticosteroids for asthma.
* History of malignancy (except patients with surgically cured basal cell or squamous cell skin cancers who will be eligible)
* History of organ transplantation
* Negative HIV-positive status determined by history at screening or known history of any other immuno-suppressing disease.
* Severe comorbidities (diabetes mellitus requiring insulin, CHF (EF<50% at baseline will be exclusionary) of any severity, MI, CVA or TIA within 3 months of screening visit, unstable angina pectoris, oxygen-dependent severe pulmonary disease
* Subject is currently enrolled in another investigational device or drug trial(s), or subject has received other investigational agent(s) within 28 days of baseline visit.
* Subjects who have known hypersensitivity to Squaric acid or any of its components.
* History of recent alcohol or substance abuse (< 1 year)
* Any condition judged by the investigator to cause this clinical trial to be detrimental to the patient.
* History of psychiatric disease that would interfere with the patient's ability to comply with the study protocol
* History of non-compliance with other therapies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra B Kimball, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.2% Squaric Acid: 0.2% Squaric Acid solution disolved in dimethyl sulfoxide will be applied
  Squaric Acid solution
- 0.5% Squaric Acid: 0.5% Squaric Acid solution disolved in dimethyl sulfoxide will be applied
  Squaric Acid solution
- Placebo Solution: Patients in placebo group will be given dimethyl sulfoxide.
  Placebo solution
Period: Overall Study
Arm/Group | 0.2% Squaric Acid | 0.5% Squaric Acid | Placebo Solution
Started | 17 | 18 | 19
Completed | 14 | 13 | 15
Not Completed | 3 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.2% Squaric Acid | 0.5% Squaric Acid | Placebo Solution | Total
Number analyzed (Participants) | 17 | 18 | 19 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 18 | 19 | 52
  >=65 years | 2 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.86 (13.68) | 47.21 (9.37) | 44.13 (10.88) | 44.93 (11.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 13 | 40
  Male | 3 | 5 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 3
  White | 13 | 17 | 18 | 48
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 19 | 54
Number of Outbreaks a year [Mean (Standard Deviation); unit: frequency per year] | 7.06 (1.71) | 7.81 (1.81) | 8.14 (2.42) | 7.68 (2.02)

OUTCOME MEASURES:

1. Primary Outcome: Subjects With at Least One Form of Contact With Study Staff With no Herpes Labialis Outbreaks Within 119 Days of Sensitization
Description: Percent of subjects with no reported herpes labialis outbreak within 119 days of sensitization over total number of subjects after one form of contact with study staff
Time Frame: 8 months
Population: Because most patients who received 2% SADBE for sensitization did not experience another herpes outbreak and thus did not receive a subsequent treatment dose, we grouped both squaric acid treatment arms together for analysis since both groups had received the same sensitization dose of 2%.
Measure: Number; unit: percentage of particpants
Groups:
- 2% Squaric Acid Sensitization: 2% Squaric Acid solution will be applied for sensitization to the inner arm.
  Squaric Acid solution
Arm/Group | 2% Squaric Acid Sensitization | Placebo Solution
Number analyzed (Participants) | 27 | 15
percentage of particpants | 62.96 | 20

2. Secondary Outcome: Number of Adverse Events Reported
Description: To assess the safety and tolerability of squaric acid solution the number of adverse events in each treatment arm will be collected and compared.
Time Frame: 8 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | 0.2% Squaric Acid | 0.5% Squaric Acid | Placebo Solution
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 9/17 | 6/18 | 3/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.2% Squaric Acid (N=17) | 0.5% Squaric Acid (N=18) | Placebo Solution (N=19)
Non Serious Itching, Redness, or Swelling (Skin and subcutaneous tissue disorders) | 8 (8) | 5 (5) | 2 (2) — Subjects who reported itching, redness, or swelling and were recorded as a non-serious AE
Other Non Serious AE (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) — Other AEs that were reported by subjects but were non-serious

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No